CLINICAL TRIAL: NCT05388565
Title: Testing the Domestic Violence Enhanced Perinatal Care in China
Brief Title: Domestic Violence Enhanced Perinatal Care Program in China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Shandong University (Other); Soochow University (Other)
Responsible Party: Principal Investigator, Yang Li, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SVRI2022
Record Dates: First submitted 2022-05-17; First posted 2022-05-24 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Intimate Partner Violence
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The DOVE in China Intervention Group (Experimental): Our intervention consists of four major components: a) information about IPV and effects on maternal and infant health, b) danger assessment, c) options and safety plan, and d) resources.
  Interventions: Behavioral: Domestic Violence Enhanced Perinatal Care Program
- The Control Group (Placebo Comparator): The control group will be provided with a standard of care including usual perinatal care (e.g., prenatal health education) and a list of resource information (e.g., crisis lines, local IPV, and mental health resources).
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Domestic Violence Enhanced Perinatal Care Program — Our intervention consists of four major components: a) information about IPV and its effects on maternal and infant health, b) danger assessment, c) options and safety plan, and d) resources.
  Arms: The DOVE in China Intervention Group
Behavioral: Standard of Care — Usual perinatal care (e.g., prenatal health education) and a list of resource information (e.g., crisis lines, local IPV and mental health resources)
  Arms: The Control Group

SUMMARY:
The proposed project addresses intimate partner violence (IPV) against pregnant women, which is a serious social and health issue. Pregnant women represent a particularly vulnerable population of IPV survivors in China, who have been largely underserved. There have been no interventions developed in China to prevent maternal IPV and its effects on maternal and infant health. The proposed project is the first structured IPV intervention integrated into prenatal care in China, which may have the potential to be translated into more prenatal clinics in China to prevent violence against pregnant women and improve maternal and infant health.

DETAILED DESCRIPTION:
Intimate partner violence (IPV) is a serious social and health issue. It is prevalent during pregnancy and in the postpartum period, causing tremendous effects on maternal and child health such as maternal depression, preterm birth, low birth weight, and impaired child neuropsychological development. However, IPV has been overlooked and is a low priority in China. No IPV intervention and prevention program has been implemented in China to help women deal with IPV in the perinatal period and eliminate its effects on maternal and child health. The Domestic Violence Enhanced Home Visitation Program (DOVE), which is a structured IPV intervention integrated into the perinatal home visitation program in the United States, focuses on educating and empowering women about IPV and their options for preventing further IPV. Building on the demonstrated effectiveness of the DOVE intervention in preventing IPV as well as the well-established perinatal care system in China, we adapted the DOVE intervention for the context of perinatal care in China. The aim of the proposed project is to test the feasibility and acceptability of the adapted DOVE intervention ("DOVE in China") in reducing maternal IPV and infant exposure to IPV and improving maternal and child health in a sample of women recruited from two perinatal clinics located in two cities (richer vs. poorer) of China. The pilot study will use a randomized two-arm pre-posttest control group design with repeated measures and mixed methods. A total of 25 women per group, who are in early pregnancy and screened positive for IPV in the year before pregnancy or during the current pregnancy, will be recruited at each of the two perinatal clinics. The intervention group will receive three prenatal sessions and one postpartum session, while the control group will receive standard of care. The frequency of IPV, depression, perceived stress, safety behaviors, birth outcomes, and child growth and development will be assessed on the web-based survey. The phone interview will ask about women's acceptability and satisfaction with the intervention and how it impacts their well-being. All women will complete the survey at baseline, 36-40 weeks before delivery, and 3 and 6 months postpartum. The interview will be conducted with women in the intervention group immediately post-intervention. The findings will help enhance the intervention by making appropriate modifications to the processes and procedures involved and provide a foundation upon which to implement a subsequent effectiveness trial. The findings will be disseminated through various means (e.g., publications, presentations). The long-term goal is to create an integrated, sustainable model for the universal screening, assessment, and treatment of IPV in China's perinatal care and improve the health of abused women and their infants.

ELIGIBILITY:
Inclusion Criteria:

* Being in early pregnancy (less than 13 weeks gestation) and screened positive for IPV in the year before pregnancy or during the current pregnancy.

Exclusion Criteria:

* Women who are not able to read and understand Chinese.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 100 (Estimated)
Dates: Start 2023-02-25 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Intimate Partner Violence | Baseline
  The Revised Conflict Tactics Scales (CTS2) will be used to measure the frequency of violent behaviors used by the partner. Higher total scores indicate more frequent violent behaviors from the partner.
Intimate Partner Violence | 36-40 weeks before delivery
  The Revised Conflict Tactics Scales (CTS2) will be used to measure the frequency of violent behaviors used by the partner. Higher total scores indicate more frequent violent behaviors from the partner.
Intimate Partner Violence | 3 months postpartum (6 weeks post-intervention)
  The Revised Conflict Tactics Scales (CTS2) will be used to measure the frequency of violent behaviors used by the partner. Higher total scores indicate more frequent violent behaviors from the partner.
Intimate Partner Violence | 6 months postpartum (18 weeks post-intervention)
  The Revised Conflict Tactics Scales (CTS2) will be used to measure the frequency of violent behaviors used by the partner. Higher total scores indicate more frequent violent behaviors from the partner.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong University, Jinan, Shandong, China